CLINICAL TRIAL: NCT02065674
Title: Therapeutic Efficacy of Homoeopathic Mother Tincture of "Abroma Agusta" in Changing the Level of Glycated Hb (HbA1c %) in Diabetes Mellitus Type II (NIDDM
Brief Title: Therapeutic Efficacy of "Abroma Agusta" in HbA1c % in NIDDM
Acronym: ABOMNIDDM
Status: Available | Type: Expanded Access
Sponsor: Fr Muller Homoeopathic Medical College (Other)
Responsible Party: Principal Investigator, dr rita chakraborty, PROFESSOR, Head of The Department of Repertory, Fr Muller Homoeopathic Medical College
Other Study IDs: ABROAGUS01
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Type II Diabetes Mellitus
Keywords: type II Diabetes mellitus; FBS; PPBS; HbA1c%
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Abroma Augusta Q (mother tincture) — 30 drops in 1 cup of water three times a day for 3 months
  Other Names: Abroma Augustum,

SUMMARY:
Objective: To ascertain whether homoeopathic medicine ABROMA AUGUSTA has a clinical role in changing the Glycated Hb Level in Diabetes mellitus Type II.

Abstract:

Background: Type 2 diabetes mellitus (T2DM) is one of the most important epidemic diseases in the world in this century, and accounts for 90% of cases of diabetes globally. Studies have suggested that Abroma Augusta plays a role in acute controlling blood glucose level. The aim of this study was to evaluate the efficacy of "Abroma Augusta Ѳ" in chronic control through GlycatedHb (HbA1c %) in Diabetes Mellitus Type 2 (NIDDM) as a pretest post-test study.

DETAILED DESCRIPTION:
Introduction:

Diabetes mellitus type 2 (noninsulin-dependent diabetes mellitus (NIDDM) or adult-onset diabetes) is a metabolic disorder that is characterized by hyperglycemia (high blood sugar) in the context of insulin resistance and relative lack of insulin. According to recent survey reports about 5% of the total world population is suffering from Diabetes Mellitus. The incidence rate is also reasonably high in India. Currently about 20% of Indian Population is at High risk to develop Diabetes Mellitus in future i.e. they are having abnormal glucose Tolerance test. Studies have revealed that diabetic women suffer more than men. Diabetes is the single most important metabolic disease which can affect nearly every organ system in the body. According to the World Health Organization estimates, India had 32 million diabetic subjects in the year 2000 and this number would increase to 80 million by the year 2030. The International Diabetes Federation (IDF) also reported that the total number of diabetic subjects in India is 41 million in 2006 and that this would rise to 70 million by the year 2025. A male who is diabetic has double the chances of heart failure. In case of women it grows to almost 5 times and it is 8 times more if the patient is a young female.

The prevalence of diabetes is rapidly rising all over the globe at an alarming rate1 . Over the past 30 yr, the status of diabetes has changed from being considered as a mild disorder of the elderly to one of the major causes of morbidity and mortality affecting the youth and middle aged people. It is important to note that the rise in prevalence is seen in all six inhabited continents of the globe2 . Although there is an increase in the prevalence of type 1 diabetes also, the major driver of the epidemic is the more common form of diabetes, namely type 2 diabetes, which accounts for more than 90 per cent of all diabetes cases. Nowhere is the diabetes epidemic more pronounced than in India as the World Health Organization (WHO) reports show that 32 million people had diabetes in the year 2000. The International Diabetes Federation (IDF) estimates the total number of diabetic subjects to be around 40.9 million in India and this is further set to rise to 69.9 million by the year 2025.

Long-term complications of diabetes develop gradually. The longer you have diabetes - and the less controlled your blood sugar - the higher the risk of complications. Eventually, diabetes complications may be disabling or even life-threatening. Possible complications include:

* Cardiovascular disease.Diabetes dramatically increases the risk of various cardiovascular problems, including coronary artery disease with chest pain (angina), heart attack, stroke and narrowing of arteries (atherosclerosis).
* Nerve damage (neuropathy). Excess sugar can injure the walls of the tiny blood vessels (capillaries) that nourish your nerves, especially in your legs. This can cause tingling, numbness, burning or pain that usually begins at the tips of the toes or fingers and gradually spreads upward. Left untreated, you could lose all sense of feeling in the affected limbs. Damage to the nerves related to digestion can cause problems with nausea, vomiting, diarrhea or constipation. For men, it may lead to erectile dysfunction.
* Kidney damage (nephropathy). The kidneys contain millions of tiny blood vessel clusters (glomeruli) that filter waste from your blood. Diabetes can damage this delicate filtering system. Severe damage can lead to kidney failure or irreversible end-stage kidney disease, which may require dialysis or a kidney transplant.
* Eye damage (retinopathy). Diabetes can damage the blood vessels of the retina (diabetic retinopathy), potentially leading to blindness. Diabetes also increases the risk of other serious vision conditions, such as cataracts and glaucoma.
* Foot damage. Nerve damage in the feet or poor blood flow to the feet increases the risk of various foot complications. Left untreated, cuts and blisters can develop serious infections, which often heal poorly. These infections may ultimately require toe, foot or leg amputation.
* Skin conditions. Diabetes may leave you more susceptible to skin problems, including bacterial and fungal infections.
* Hearing impairment. Hearing problems are more common in people with diabetes.
* Alzheimer's disease. Type 2 diabetes may increase the risk of Alzheimer's disease. The poorer your blood sugar control, the greater the risk appears to be. Although there are theories as to how these disorders might be connected, none has yet been proved.

So Diabetes is associated with long term complications that affect almost every major part of the body. Type 2 diabetes is initially managed by increasing exercise and dietary changes. If blood sugar levels are not adequately lowered by these measures, medications or intervention is needed. In those on medication, there is absolute requirement of routinely check up of blood sugar levels.

There is good number of Homoeopathic medicine to control blood sugar level. They are Cephalandra Indica, Syzegium, Gymnema Sylvestree, Abroma Augusta, Rhus Aromatica rtc. It is noticed that the blood sugar (HbA1c) is not controlled by other system of medicine; the patients come for Homoeopathic treatment and after homoeopathic treatment there is a remarkable improvement in FBS, PPBS as well as HbA1c along with the general improvement of health like tiredness, lethargy, numbness, polyurea, polydypsia and polyphagia etc. But there is no scientific validation for that. Among those Abroma Augusta is selected for this study and this study is conducted for achieving the scientific validation, the homoeopathic hypoglycemic "Abroma Augusta".

ABROMA AUGUSTA Family: Sterculiaceae Bengali/vernacular name: Ulatkambal. Tribal name: Polumaoeba (Chakma); Daiya (Garo). English name: Devil's Cotton. Usually it has been used widely as an emmenagogue but its glycemic use is rare. Abroma Augusta commonly known as Olat Kambal. The plant of Abroma Augusta grows wild throughout the hotter part of India. In ancient times, it was used therapeutically as an emmenagogue in menstrual disorders. Late Dr. D.N.Roy of Calcutta proved this drug. A tincture of the drug is prepared from its leaves according to class III of American Homeopathic Pharmacopoea. It is used in diabetes insipidus with very gratifying results. Clinically it is indicated in Diabetes, albuminuria, enuresis, debility, vertigo, sleeplessness, carbuncle, amenorrhoea and dysmenorrhoea.

Description of the plant: ABROMA AUGUSTA L. is a large shrub. Leaves large, 10-15 by 10-12.5 cm, repand - denticulate, upper smaller, narrower, entire. Flower is solitary, auxiliary, pendulous, peduncle up to 4 cm long; sepals 2.5 cm, lanceolate; petals scarcely exceeding the sepals, dark red.

Chemical constituents:

Leaves contain taraxerol, its acetate and β-sitosterol. Stem bark contains friedelin and β-sitosterol. Root and root bark contain gum, fixed oil, resin, alkaloids, abromine, choline and betaine, β-sitosterol, stigmasterol, digitonide, magenesium salts of hydroxyl acids and polysaccharide. Seeds contain 20.2% fixed oil with 71.5% linoleic acid. Augustic acid an oleanane derivative and a stigmasterol glycoside have been isolated from the roots. Heartwood contains β-sitosterol, glycol and octacosane-1, 28-diol (Ghani, 2003; Rastogi & Mehrotra, 1993; Asolkar et al., 1992). Among them Taraxerol is the most important component which has hypoglycemic as well as anti-inflammatory action. It also contains flavinoid & phenolic component and they are phyto- antioxidant.

Homoeopathic uses: Fragmentary proving was conducted by Dr. D.N. Ray of Calcutta in 1919 and Dr. Jugal Kishore of New Delhi in 1972. It has been subsequently proved by CCRH and has shown its affinity for female reproductive organs producing symptoms of dysmenorrhoea and leucorrhoea, which have been confirmed during verification trials too.

Diabetes mellitus - Urine profuse < at night and of high specific gravity. Excessive thirst with dryness of mouth. Patient suffers from insomnia and prostration, and patient is averse to do any physical and intellectual labour. Mentally patient is of irritable nature, forgetful and morose.

Dysmenorrhoea - Colicky pains in lower abdomen. Menses are irregular, lasting for short or long time. Blood is dark and clotted.

There is lots of study on Aboma Augusta in modern system of Medicie as well as the Ayurveda on Rats and it was proved that this drug has not only the hypoglycemic effect (Taraxerol) but also has effect on antioxidant and lipid control. So this study was conducted to investigate the therapeutic efficacy on Human being.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria Age 30 Years above Both Sexes NIDDM FBS - 110-300mg/dl HbA1c above ≤ 6.5

-

Exclusion Criteria:

* Patient with major complications like diabetic retinopathy and cardiomyopathy. IDDM HbA1c above 11%

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2014-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: dr rita chakraborty, MD, Principal Investigator — Fr Muller Homoeopathic Medical College
Locations (1):
- ,Father Muller Homoeopathic Medical College, Prasanth Nivas Ashram Nmpt Hospital, Mangalore, Karnataka, India